CLINICAL TRIAL: NCT02733380
Title: The Efficacy and Safety of Chidamide Combined With VDDT Regimen（Vinorelbine，Liposomal Doxorubicin，Dexamethasone and Thalidomide） in Relapse and Refractory Patients With Diffuse Large B Cell Lymphoma
Brief Title: Chidamide Combined With VDDT Regimen in the Relapse and Refractory Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYML-01
Record Dates: First submitted 2016-03-25; First posted 2016-04-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2018-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Relapsed and refractory; Histone deacetylase inhibitor; Chidamide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Vinorelbine; liposomal doxorubicin; Mitoxantrone; Dexamethasone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide combined with VDDT regimen (Experimental): Chidamide 30mg，Oral twice a week with an interval of no less than 3 days combined with regimen：VDDT（Vinorelbine，Liposomal doxorubicin or mitoxantrone ，Dexamethasone and Thalidomide）：repeated every 14 days ，up to 12 cycles
  Interventions: Drug: Chidamide; Drug: Vinorelbine; Drug: Liposomal Doxorubicin or mitoxantrone; Drug: Dexamethasone; Drug: Thalidomide

INTERVENTIONS:
Drug: Chidamide — 30mg , Oral twice a week(with an interval of no less than 3 days,;e.g. Monday and Thursday，Tuesday and Friday) until disease progression or unacceptable toxicity develops
Drug: Vinorelbine — 20mg/m2， IV on day 1 of each 14 day cycle until disease progression or unacceptable toxicity develops, up to 12 cycles
Drug: Liposomal Doxorubicin or mitoxantrone — 20mg/m2, IV on day 1 of each 14 day cycle（Note：for patients who can not afford the liposomal doxorubicin，may be replaced into mitoxantrone 8mg/m2, IV on day1 of each 14 day cycle） until disease progression or unacceptable toxicity develops, up to 12 cycles
Drug: Dexamethasone — 10mg/m2 , IV on day 1-5 of each 14 day cycle until disease progression or unacceptable toxicity develops, up to 12 cycles
Drug: Thalidomide — 100mg,Oral at night on each day until disease progression or unacceptable toxicity develops, up to 24 weeks

SUMMARY:
This is a prospective phase II clinical trial to observe the efficacy and safety of Chidamide combined with VDDT(vinorelbine，liposomal doxorubicin，dexamethasone and thalidomide) in relapsed and refractory patients with diffuse large B-cell lymphoma(DLBCL).

DETAILED DESCRIPTION:
There are one third of diffuse large B-cell Lymphoma patients suffering relapse and refractory, which are the major cause of death among these patients. Vinorelbine，liposomal doxorubicin，mitoxantrone, dexamethasone and thalidomide have been used in the therapy of patients who failed with Second-line treatments in our center. This regimen is well tolerated but the effect needs to be improved. Chidamide，a histone deacetylase inhibitor has been approved for the treatment of refractory T-cell lymphoma in China. The goal is to assess the efficacy and safety of chidamide combined with VDDT（vinorelbine，liposomal doxorubicin，dexamethasone and thalidomide） in relapse and refractory patients with diffuse large B-cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as diffuse large B-cell Lymphoma based on the 2008 WHO classification of tumors of haematopoietic and lymphoid tissues
2. Failed with second-line therapy
3. Having at least one measurable lesions
4. Age between 18 to 75 years old
5. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-1
6. Neutrophils more than 1.5*10^9/L; Platelets more than 90*10^9/L Hemoglobin: more than 90g/L.
7. Life expectancy no less than 3 months
8. No receiving chemotherapy in 4 weeks before enrollment
9. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Pregnant ，lactating and patients at reproductive age who refuse to practice contraception
2. QTc prolonging >450ms，ventricular tachycardia，atrial fibrillation，cardiac conduction block， myocardial infarction in less than 1 year， congestive heart failure，coronary heart disease which needs medication.
3. Organ transplant recipients
4. Active bleeding
5. Thrombus，embolism，cerebral hemorrhage，cerebral infarction
6. Important organ operation in less than 6 weeks
7. Abnormal liver function（Note：total bilirubin >1.5 times the upper limit of normal，AST or ALT >2.5 times the upper limit of normal （Note：5 times the upper limit of normal for patients with liver involvement）），abnormal renal function（Note：serum creatinine >1.5 times the upper limit of normal），fluid and electrolyte disorders
8. Mental illness or unable to sign the informed consent
9. Drug addiction history or alcoholism which may interfere the experimental results.
10. Researchers determine unsuited to participate in this trial
11. Known allergy to any kind of study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
objective response rate | every 8 weeks until 1 year after last patient's enrollment
  the total proportion of patients with complete response（CR or CRu）and partial response（PR）
adverse events | from the date of first cycle of treatment to 1 year after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
abnormal laboratory examinations | from the date of first enrollment to 1 year after last patient's enrollment
  includes type, incidence, relationship with treatment and severity of abnormal laboratory examinations.
incidence and relationship with study drugs of grade 3-4 adverse events and abnormal laboratory examinations | from the date of first cycle of treatment to 1 year after last patient's enrollment
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03) and abnormal laboratory examinations

SECONDARY OUTCOMES:
progression-free survival | from the day of treatment to the date of first documented progression，up to 1 year after last patient's enrollment
  from date of first day of treatment to the date of first documented
duration of response | from the day of first documented response to first documented progression or death，up to 1 year after last patient's enrollment
  from the first day of documented response to disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

REFERENCES:
- [Result] Wynder EL. Listen to nature. The challenge of lifestyle medicine. Soz Praventivmed. 1991;36(3):137-46. doi: 10.1007/BF01352692. PMID 1950172
- [Result] Witt O, Deubzer HE, Milde T, Oehme I. HDAC family: What are the cancer relevant targets? Cancer Lett. 2009 May 8;277(1):8-21. doi: 10.1016/j.canlet.2008.08.016. Epub 2008 Sep 27. PMID 18824292
- [Result] Khan AN, Tomasi TB. Histone deacetylase regulation of immune gene expression in tumor cells. Immunol Res. 2008;40(2):164-78. doi: 10.1007/s12026-007-0085-0. PMID 18213528
- [Result] Pasqualucci L, Dominguez-Sola D, Chiarenza A, Fabbri G, Grunn A, Trifonov V, Kasper LH, Lerach S, Tang H, Ma J, Rossi D, Chadburn A, Murty VV, Mullighan CG, Gaidano G, Rabadan R, Brindle PK, Dalla-Favera R. Inactivating mutations of acetyltransferase genes in B-cell lymphoma. Nature. 2011 Mar 10;471(7337):189-95. doi: 10.1038/nature09730. PMID 21390126
- [Result] Morin RD, Mendez-Lago M, Mungall AJ, Goya R, Mungall KL, Corbett RD, Johnson NA, Severson TM, Chiu R, Field M, Jackman S, Krzywinski M, Scott DW, Trinh DL, Tamura-Wells J, Li S, Firme MR, Rogic S, Griffith M, Chan S, Yakovenko O, Meyer IM, Zhao EY, Smailus D, Moksa M, Chittaranjan S, Rimsza L, Brooks-Wilson A, Spinelli JJ, Ben-Neriah S, Meissner B, Woolcock B, Boyle M, McDonald H, Tam A, Zhao Y, Delaney A, Zeng T, Tse K, Butterfield Y, Birol I, Holt R, Schein J, Horsman DE, Moore R, Jones SJ, Connors JM, Hirst M, Gascoyne RD, Marra MA. Frequent mutation of histone-modifying genes in non-Hodgkin lymphoma. Nature. 2011 Jul 27;476(7360):298-303. doi: 10.1038/nature10351. PMID 21796119
- [Result] Mondello P, Younes A. Emerging drugs for diffuse large B-cell lymphoma. Expert Rev Anticancer Ther. 2015 Apr;15(4):439-51. doi: 10.1586/14737140.2015.1009042. Epub 2015 Feb 5. PMID 25652253
- [Result] Dong M, Ning ZQ, Xing PY, Xu JL, Cao HX, Dou GF, Meng ZY, Shi YK, Lu XP, Feng FY. Phase I study of chidamide (CS055/HBI-8000), a new histone deacetylase inhibitor, in patients with advanced solid tumors and lymphomas. Cancer Chemother Pharmacol. 2012 Jun;69(6):1413-22. doi: 10.1007/s00280-012-1847-5. Epub 2012 Feb 24. PMID 22362161
- [Result] Ning ZQ, Li ZB, Newman MJ, Shan S, Wang XH, Pan DS, Zhang J, Dong M, Du X, Lu XP. Chidamide (CS055/HBI-8000): a new histone deacetylase inhibitor of the benzamide class with antitumor activity and the ability to enhance immune cell-mediated tumor cell cytotoxicity. Cancer Chemother Pharmacol. 2012 Apr;69(4):901-9. doi: 10.1007/s00280-011-1766-x. Epub 2011 Nov 12. PMID 22080169
- [Result] Gong K, Xie J, Yi H, Li W. CS055 (Chidamide/HBI-8000), a novel histone deacetylase inhibitor, induces G1 arrest, ROS-dependent apoptosis and differentiation in human leukaemia cells. Biochem J. 2012 May 1;443(3):735-46. doi: 10.1042/BJ20111685. PMID 22339555
- [Result] Zhou Y, Pan DS, Shan S, Zhu JZ, Zhang K, Yue XP, Nie LP, Wan J, Lu XP, Zhang W, Ning ZQ. Non-toxic dose chidamide synergistically enhances platinum-induced DNA damage responses and apoptosis in Non-Small-Cell lung cancer cells. Biomed Pharmacother. 2014 May;68(4):483-91. doi: 10.1016/j.biopha.2014.03.011. Epub 2014 Mar 18. PMID 24721323
- [Result] Frys S, Simons Z, Hu Q, Barth MJ, Gu JJ, Mavis C, Skitzki J, Song L, Czuczman MS, Hernandez-Ilizaliturri FJ. Entinostat, a novel histone deacetylase inhibitor is active in B-cell lymphoma and enhances the anti-tumour activity of rituximab and chemotherapy agents. Br J Haematol. 2015 May;169(4):506-19. doi: 10.1111/bjh.13318. Epub 2015 Feb 23. PMID 25712263
- [Result] Shimizu R, Kikuchi J, Wada T, Ozawa K, Kano Y, Furukawa Y. HDAC inhibitors augment cytotoxic activity of rituximab by upregulating CD20 expression on lymphoma cells. Leukemia. 2010 Oct;24(10):1760-8. doi: 10.1038/leu.2010.157. Epub 2010 Aug 5. PMID 20686505